CLINICAL TRIAL: NCT05316701
Title: A Randomized Phase III Trial of Patients With Advanced Hematologic Malignancies Undergoing Allogeneic Hematopoietic Cell Transplantation With Either Orca-T, a T-cell-Depleted Graft With Additional Infusion of Conventional T Cells and Regulatory T Cells, or Standard-of-Care Allogeneic Graft
Brief Title: Precision-T: A Randomized Study of Orca-T in Recipients Undergoing Allogeneic Transplantation for Hematologic Malignancies
Acronym: Orca-T
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Orca Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Precision-T (PhIII component)
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Results first posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoid Leukemia; Mixed Phenotype Acute Leukemia; Undifferentiated Leukemia; Myelodysplastic Syndrome; Acute Leukemia; Therapy-Related Myelodysplastic Syndrome
Keywords: hematopoietic stem cell transplantation; acute leukemia; Myelodysplastic syndromes; matched related donor; matched unrelated donor; myelodysplastic syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Myelodysplastic Syndromes | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The Phase III is a randomized, open-label, multicenter study comparing outcomes between patients receiving Orca-T followed by single-agent tacrolimus or standard-of-care (SOC) control followed by dual agent, tacrolimus-based Graft-versus-Host-Disease (GVHD) prophylaxis regimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orca-T (Experimental): For patients randomized to the Orca-T arm, Orca-T will be administered after myeloablative conditioning regimen. Single-agent GVHD prophylaxis with tacrolimus will be administered following Tcon infusion (generally Day +3).
  Interventions: Biological: Orca-T
- Standard of Care alloHCT Control (Active Comparator): For patients randomized to the standard-of-care control arm, an unmanipulated allograft derived from the peripheral blood of a matched donor will be administered after a myeloablative conditioning regimen. Dual-agent prophylaxis consisting of tacrolimus plus methotrexate will be administered starting on Day -3.
  Interventions: Biological: Standard-of-Care

INTERVENTIONS:
Biological: Orca-T — an allogeneic stem cell and T-cell immunotherapy biologic
  Arms: Orca-T
Biological: Standard-of-Care — unmanipulated donor allograft
  Other Names: SOC
  Arms: Standard of Care alloHCT Control

SUMMARY:
This study will evaluate the safety, tolerability, and efficacy of Orca-T, an allogeneic stem cell and T-cell immunotherapy biologic manufactured for each patient (transplant recipient) from the mobilized peripheral blood of a specific, unique donor. It is composed of purified hematopoietic stem and progenitor cells (HSPCs), purified regulatory T cells (Tregs), and conventional T cells (Tcons) in participants undergoing myeloablative allogeneic hematopoietic cell transplant transplantation for hematologic malignancies.

This posting represents the Phase III component of Precision-T. The Precision-T Ph1b component is described under NCT04013685.

DETAILED DESCRIPTION:
Cross reference NCT04013685

ELIGIBILITY:
Key Inclusion Criteria:

* Matched to a related or unrelated donor who is an 8/8 match for HLA-A, -B, -C, and DRB1
* Diagnosed with one of the following diseases:

  * Acute myeloid, lymphoid or mixed phenotype leukemia in complete remission (CR) or CR with incomplete hematologic recovery (CRi), with or without the presence of known minimal residual disease
  * Myelodysplastic syndromes (MDS) that are indicated for alloHSCT per 2017 International Expert Panel recommendations and/or have therapy-related/secondary MDS, with ≤ 10% blast burden in the bone marrow
* Planned to undergo MA-alloHCT including one of the following myeloablative conditioning regimens:

  * TBI/Cy
  * TBI/Etoposide
  * BFT
* Cardiac ejection fraction at rest ≥ 45% or shortening fraction of ≥ 27% by echocardiogram or radionuclide scan (MUGA)
* Diffusing capacity of the lung for carbon monoxide (DLCO) (adjusted for hemoglobin) ≥ 50%
* Negative serum or urine beta-HCG test in females of childbearing potential
* ALT/AST < 3 times ULN
* Recipients in screening must screen negative for SARS-CoV-2 RNA using a PCR-based test
* Disease Risk Index (DRI) overall risk categorization of intermediate or high
* Total bilirubin ≤ upper limit of normal (ULN)
* Estimated glomerular filtration rate (eGFR) ≥ 60 mL/minute

Key Exclusion Criteria:

* Prior allogeneic HCT
* Currently receiving corticosteroids or other immunosuppressive therapy. Topical corticosteroids or oral systemic corticosteroid doses less than or equal to 10 mg/day are allowed.
* Planned donor lymphocyte infusion (DLI)
* Planned pharmaceutical in vivo or ex vivo T cell depletion
* Recipient positive anti-donor HLA antibodies against a mismatched allele in the selected donor
* Karnofsky performance score < 70%
* Hematopoietic cell transplantation-specific Comorbidity Index (HCT-CI) > 4
* Uncontrolled bacterial, viral or fungal infections at time of enrollment
* Seropositive for HIV-1 or -2, HTLV-1 or -2, Hepatitis B sAg, Hepatitis C antibody
* Known allergy or hypersensitivity to, or intolerance of, tacrolimus
* Documented allergy or hypersensitivity to iron dextran or bovine, murine, algal or Streptomyces avidinii proteins
* Any uncontrolled autoimmune disease requiring active immunosuppressive treatment
* Concurrent malignancies or active disease within 1 year, except non-melanoma skin cancers that have been curatively resected
* Psychosocial circumstances that preclude the patient being able to go through transplant or participate responsibly in follow up care
* Women who are pregnant or breastfeeding
* Women of childbearing potential (WOCBP) or men who have sexual contact with WOCBP unwilling to use effective forms of birth control or abstinence for one year after transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2026-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - City of Hope, Duarte, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UC Davis, Sacramento, California
  - Stanford Health Care, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Miami Hospital and Clinics - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Health System - Michigan Medicine, Ann Arbor, Michigan
  - Weill Cornell Medicine - New York-Presbyterian Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health & Sciences University - Knight Cancer Institute, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meyer E, Salhotra A, Gandhi A, Pantin J, Patel SS, Hoeg RT, Gomez-Arteaga A, Faramand RG, Tamari R, Waller EK, Kosuri S, Jimenez Jimenez AM, Holter-Chakrabarty J, Dholaria B, Chen YB, Hamilton BK, Magenau JM, Eghtedar A, Murray JM, Pavlova A, Fernhoff NB, McClellan JS, Killian S, Li A, Negrin RS, Oliai C. Orca-T versus allogeneic hematopoietic stem cell transplantation (PRECISION-T): a multicenter, randomized phase 3 trial. Blood. 2025 Dec 12:blood.2025031313. doi: 10.1182/blood.2025031313. Online ahead of print. PMID 41385341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 187 participants were randomized to treatment from 19 study centers, of which 182 participants were treated
Groups:
- Orca-T: Orca-T administered after myeloablative conditioning followed by single-agent tacrolimus
- Standard of Care: Unmanipulated allograft from peripheral blood of a matched donor after myeloablative conditioning followed by tacrolimus and methotrexate
Period: Overall Study
Arm/Group | Orca-T | Standard of Care
Started | 93 | 94
Participants Treated | 88 | 94
Completed | 0 | 2
Not Completed | 93 | 92
Not completed — Adverse Event | 0 | 1
Not completed — Death | 3 | 9
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 4
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Progression/Relapse | 14 | 9
Not completed — Received Standard of Care | 1 | 0
Not completed — Ongoing | 70 | 64

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT): All enrolled participants who were randomized to either Orca-T or standard of care (SoC), regardless of whether they received Orca-T/SoC or not; participants were analyzed according to their randomized treatment assignment
Groups:
- Total: Total of all reporting groups
Arm/Group | Orca-T | Standard of Care | Total
Number analyzed (Participants) | 93 | 94 | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 93 | 94 | 187
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 44 | 84
  Male | 53 | 50 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 24 | 50
  Not Hispanic or Latino | 62 | 59 | 121
  Unknown or Not Reported | 5 | 11 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 10 | 8 | 18
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 1 | 2 | 3
  White | 76 | 63 | 139
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 18 | 22
Region of Enrollment [Number; unit: participants]
  United States | 93 | 94 | 187
Primary Disease [Count of Participants; unit: Participants] — Primary disease at enrollment
  Participants
    Acute Lymphoid Leukemia (ALL) | 30 | 27 | 57
    Acute Myeloid Leukemia (AML) | 49 | 51 | 100
    High-risk Myelodysplastic Syndrome (MDS) | 12 | 11 | 23
    Mixed Phenotype Acute Leukemia (MPAL) | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Event-free at 12 Months for Moderate or Severe Chronic Graft-versus-Host-Disease-free Survival (cGFS) Per Endpoint Adjudication Committee (EAC)
Description: Event-free rate estimated at 12 months for cGFS per EAC, which is defined as the time from date of allogeneic hematopoietic cell transplantation (alloHCT) (ie, day 0) to date of death from any cause or first onset of moderate or severe chronic graft-versus-host disease (cGVHD) (graded per NIH consensus criteria), whichever was earliest, within 2 years after day 0. cGVHD was assessed and graded by EAC blinded to treatment assignment.
  Each participant in the study is followed for up to 730 days after transplant. Primary analysis was event driven (ie, when 56 participants had died or had moderate or severe cGVHD) and was not based on duration of follow-up. The analysis was conducted using all available data at the time that the 56th event occurred, and event-free rate at 12 months was estimated regardless of length of follow-up for individual participants. At the time of analysis, not all participants have reached 730 days of follow-up because they enrolled at different times.
Time Frame: Day 0 through 730 days after transplantation
Population: ITT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Orca-T | Standard of Care
Number analyzed (Participants) | 93 | 94
Percentage of participants | 78.0 [65.0 to 86.6] | 38.4 [26.2 to 50.5]
Statistical Analysis 1: Comparison: Orca-T vs Standard of Care; Log-rank test was stratified by randomization stratification factors; Test type: Superiority; p < 0.00001, Log Rank; Hazard Ratio (HR) = 0.26, 95% CI 2-sided [0.14 to 0.47]

2. Secondary Outcome: Event Rate at 12 Months for Time to Moderate or Severe cGVHD Per EAC
Description: Event rate estimated at 12 months for time from alloHCT to first onset of moderate or severe cGVHD defined by NIH consensus criteria within 2 years after day 0. Death within 2 years after day 0 without prior moderate or severe cGVHD was considered a competing event. cGVHD was assessed and graded by an independent EAC.
  Each participant in the study is followed for up to 730 days after transplant. The primary analysis was triggered by the 56th cGFS event (ie, when 56 participants had died or had moderate or severe chronic GVHD) and was not based on the duration of follow-up. Therefore, the analysis was conducted using all available data at the time that the 56th cGFS event occurred, and the event rate of moderate or severe cGVHD at 12 months was estimated regardless of the length of follow-up for individual participants. At the time of analysis, not all participants have reached 730 days of follow-up because they enrolled at different times.
Time Frame: Day 0 through 730 days after transplantation
Population: ITT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Orca-T | Standard of Care
Number analyzed (Participants) | 93 | 94
Percentage of participants | 12.6 [5.3 to 23.1] | 44.0 [31.3 to 56.1]
Statistical Analysis 1: Comparison: Orca-T vs Standard of Care; Gray's test was stratified by randomization stratification factors; Test type: Superiority; p = 0.00002, Gray's test; Hazard Ratio (HR) = 0.19, 95% CI 2-sided [0.08 to 0.43]

3. Secondary Outcome: Event-free at 12 Months for Overall Survival (OS)
Description: Event-free rate estimated at 12 months for OS, which is defined as time from randomization to death from any cause.
  Each participant in the study is followed for up to 730 days after transplant. The analysis was triggered by the 56th cGFS event (ie, when 56 participants had died or had moderate or severe chronic GVHD) and was not based on the duration of follow-up. Therefore, the analysis was conducted using all available data at the time that the 56th cGFS event occurred, and the event-free rate of OS at 12 months was estimated regardless of the length of follow-up for individual participants. At the time of analysis, not all participants have reached 730 days of follow-up because they enrolled at different times.
Time Frame: Up to 730 days after end of enrollment
Population: ITT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Orca-T | Standard of Care
Number analyzed (Participants) | 93 | 94
Percentage of participants | 93.9 [85.8 to 97.4] | 83.1 [72.9 to 89.8]
Statistical Analysis 1: Comparison: Orca-T vs Standard of Care; Log-rank test was stratified by randomization stratification factors; Test type: Superiority; p = 0.11823, Log Rank; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.20 to 1.22]

4. Secondary Outcome: Event-free Rate at 12 Months for Graft-versus-host Disease-free and Relapse-free Survival (GRFS) Per EAC
Description: Event-free rate estimated at 12 months for GRFS, which is defined as time from alloHCT to death from any cause, relapse, the first onset of grade 3 or 4 acute GVHD (graded per Mount Sinai aGVHD International Consortium [MAGIC] criteria), or the first onset of moderate or severe cGVHD (graded per NIH consensus criteria), whichever is earliest, within 2 years from day 0 as assessed by independent EAC.
  Each participant in the study is followed for up to 730 days after transplant. The analysis was triggered by the 56th cGFS event (ie, when 56 participants had died or had moderate or severe cGVHD) and not based on duration of follow-up. Therefore, analysis was conducted using all available data at the time that the 56th cGFS event occurred, and event-free rate of GRFS at 12 months was estimated regardless of length of follow-up for individual participants. At time of analysis, not all participants have reached 730 days of follow-up because they enrolled at different times.
Time Frame: Day 0 through 730 days after transplantation
Population: ITT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Orca-T | Standard of Care
Number analyzed (Participants) | 93 | 94
Percentage of participants | 63.1 [50.0 to 73.6] | 30.9 [20.0 to 42.4]
Statistical Analysis 1: Comparison: Orca-T vs Standard of Care; Log-rank test was stratified by randomization stratification factors; Test type: Superiority; p = 0.00003, Log Rank; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.23 to 0.60]

ADVERSE EVENTS:
Time Frame: A treatment-emergent AE (TEAE) was any AE that started on or after alloHCT infusion (Orca-T or SoC) through study completion (day +730).
Description: Safety Analysis Set: Participants in the ITT analysis set who received either Orca-T or SoC, analyzed according to treatment received
Arm/Group | Orca-T | Standard of Care
All-Cause Mortality (participants affected / at risk) | 3/88 | 9/94
Serious Adverse Events (participants affected / at risk) | 34/88 | 53/94
Other Adverse Events (participants affected / at risk) | 88/88 | 94/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Orca-T (N=88) | Standard of Care (N=94)
Sepsis (Infections and infestations) | 7 | 6
Bacterial sepsis (Infections and infestations) | 4 | 4
Pneumonia (Infections and infestations) | 1 | 6
COVID-19 (Infections and infestations) | 0 | 5
Septic shock (Infections and infestations) | 1 | 3
Staphylococcal sepsis (Infections and infestations) | 1 | 3
Adenovirus infection (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 1 | 1
Rhinovirus infection (Infections and infestations) | 1 | 1
BK virus infection (Infections and infestations) | 0 | 1
Cellulitis orbital (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Cystitis viral (Infections and infestations) | 0 | 1
Cytomegalovirus colitis (Infections and infestations) | 0 | 1
Cytomegalovirus enterocolitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Fungaemia (Infections and infestations) | 0 | 1
Metapneumovirus infection (Infections and infestations) | 1 | 0
Mycobacterium chelonae infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Nocardiosis (Infections and infestations) | 0 | 1
Norovirus infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 1
Pneumonia escherichia (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Sapovirus infection (Infections and infestations) | 0 | 1
Shigella infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Viraemia (Infections and infestations) | 1 | 0
Viral haemorrhagic cystitis (Infections and infestations) | 1 | 0
Acute graft-versus-host disease (Immune system disorders) | 6 | 12
Chronic graft-versus-host disease (Immune system disorders) | 1 | 6
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 3
Mucosal inflammation (General disorders) | 0 | 3
Hypotension (Vascular disorders) | 0 | 3
Distributive shock (Vascular disorders) | 1 | 1
Embolism (Vascular disorders) | 0 | 2
Hypovolaemic shock (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Venous occlusion (Vascular disorders) | 0 | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 3 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Acute cholecystitis necrotic (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 4
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Uraemic encephalopathy (Nervous system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Aortic injury (Injury, poisoning and procedural complications) | 0 | 1
Transplant failure (Injury, poisoning and procedural complications) | 1 | 0
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Orca-T (N=88) | Standard of Care (N=94)
Nausea (Gastrointestinal disorders) | 79 | 79
Diarrhoea (Gastrointestinal disorders) | 71 | 83
Vomiting (Gastrointestinal disorders) | 43 | 43
Stomatitis (Gastrointestinal disorders) | 32 | 50
Constipation (Gastrointestinal disorders) | 26 | 35
Abdominal pain (Gastrointestinal disorders) | 27 | 32
Dyspepsia (Gastrointestinal disorders) | 21 | 31
Dry mouth (Gastrointestinal disorders) | 19 | 15
Oesophagitis (Gastrointestinal disorders) | 11 | 12
Haemorrhoids (Gastrointestinal disorders) | 12 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 9
Proctalgia (Gastrointestinal disorders) | 7 | 6
Abdominal pain upper (Gastrointestinal disorders) | 4 | 9
Abdominal distension (Gastrointestinal disorders) | 7 | 5
Dysphagia (Gastrointestinal disorders) | 4 | 7
Oral pain (Gastrointestinal disorders) | 5 | 5
Colitis (Gastrointestinal disorders) | 1 | 5
Flatulance (Gastrointestinal disorders) | 6 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 49 | 53
Hypokalaemia (Metabolism and nutrition disorders) | 18 | 24
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 23
Hyponatraemia (Metabolism and nutrition disorders) | 15 | 12
Vitamin D deficiency (Metabolism and nutrition disorders) | 9 | 17
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 13
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 12
Dehydration (Metabolism and nutrition disorders) | 5 | 6
Hypervolaemia (Metabolism and nutrition disorders) | 4 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 5
Hypophagia (Metabolism and nutrition disorders) | 1 | 5
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 5
Fatigue (General disorders) | 50 | 48
Mucosal inflammation (General disorders) | 29 | 26
Oedema peripheral (General disorders) | 21 | 26
Pyrexia (General disorders) | 20 | 22
Pain (General disorders) | 4 | 10
Chills (General disorders) | 8 | 4
Oedema (General disorders) | 4 | 7
Non-cardiac chest pain (General disorders) | 6 | 4
Chest pain (General disorders) | 1 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 46 | 44
Febrile neutropenia (Blood and lymphatic system disorders) | 32 | 42
Anaemia (Blood and lymphatic system disorders) | 36 | 34
Neutropenia (Blood and lymphatic system disorders) | 25 | 25
Leukopenia (Blood and lymphatic system disorders) | 22 | 16
Lymphopenia (Blood and lymphatic system disorders) | 6 | 5
Eosinophilia (Blood and lymphatic system disorders) | 0 | 6
Sepsis (Infections and infestations) | 5 | 3
COVID-19 (Infections and infestations) | 7 | 6
Candida infection (Infections and infestations) | 7 | 9
Oral candidiasis (Infections and infestations) | 4 | 9
BK virus infection (Infections and infestations) | 4 | 7
Pneumonia (Infections and infestations) | 0 | 5
Rhinovirus infection (Infections and infestations) | 3 | 7
Folliculitis (Infections and infestations) | 5 | 6
Cytomegalovirus infection reactivation (Infections and infestations) | 6 | 4
Conjunctivitis (Infections and infestations) | 1 | 7
Skin infection (Infections and infestations) | 1 | 6
Headache (Nervous system disorders) | 33 | 39
Tremor (Nervous system disorders) | 12 | 19
Dizziness (Nervous system disorders) | 15 | 15
Dysgeusia (Nervous system disorders) | 14 | 11
Neuropathy peripheral (Nervous system disorders) | 8 | 7
Paraesthesia (Nervous system disorders) | 5 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 23 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 23
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 10
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 18
Rash (Skin and subcutaneous tissue disorders) | 14 | 17
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 9
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 11 | 13
Erythema (Skin and subcutaneous tissue disorders) | 10 | 10
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 10
Dermatitis (Skin and subcutaneous tissue disorders) | 7 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 1
Acute graft-versus-host disease (Immune system disorders) | 25 | 33
Chronic graft-versus-host disease (Immune system disorders) | 13 | 40
Hypogammaglobulinaemia (Immune system disorders) | 3 | 5
Blood creatinine increased (Investigations) | 23 | 22
Alanine aminotransferase increased (Investigations) | 13 | 15
Aspartate aminotransferase increased (Investigations) | 10 | 13
Weight decreased (Investigations) | 9 | 7
Blood bilirubin increased (Investigations) | 5 | 10
Blood alkaline phosphatase increased (Investigations) | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Insomnia (Psychiatric disorders) | 25 | 32
Anxiety (Psychiatric disorders) | 8 | 13
Confusional state (Psychiatric disorders) | 1 | 5
Hypertension (Vascular disorders) | 20 | 19
Hypotension (Vascular disorders) | 13 | 10
Orthostatic hypotension (Vascular disorders) | 4 | 6
Sinus tachycardia (Cardiac disorders) | 15 | 21
Tachycardia (Cardiac disorders) | 3 | 10
Dry eye (Eye disorders) | 6 | 8
Vision blurred (Eye disorders) | 8 | 6
Haematuria (Eye disorders) | 6 | 10
Dysuria (Eye disorders) | 9 | 4
Pollakiuria (Eye disorders) | 6 | 5
Hypertransaminasaemia (Hepatobiliary disorders) | 13 | 10
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 6
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 8
Decreased appetite (Metabolism and nutrition disorders) | 40 | 47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT05316701/Prot_SAP_000.pdf